CLINICAL TRIAL: NCT01325597
Title: Effects of Functional Electrical Stimulation and Inspiratory Muscle Training in Heart Failure Patients: Randomized Clinical Trial
Brief Title: Effects of Functional Electrical Stimulation and Inspiratory Muscle Training in Heart Failure Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Graciele Sbruzzi, Doutora, Instituto de Cardiologia do Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UP 4546/10
Record Dates: First submitted 2011-03-14; First posted 2011-03-30 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Heart Failure
Keywords: Heart failure; Electric stimulation; Breathing exercises
MeSH Terms: conditions — Heart Failure | interventions — Electric Stimulation; Breathing Exercises; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Combined training (Experimental): Training with functional electrical stimulation added by inspiratory muscle training.
  Interventions: Other: Electrical stimulation; Other: Inspiratory muscle training; Other: Control group
- Electrical stimulation (Experimental): FES will be applied at 15 Hz, 0.4 ms pulse width, 10-s contraction time, 50-s resting time and maximum tolerable intensity, 3 sessions per week, for 12 weeks
  Interventions: Other: Combined training; Other: Inspiratory muscle training; Other: Control group
- Inspiratory muscle training (Experimental): IMT will be performed for 12 weeks, 5 sessions per week, with an intensity of 30% of maximal inspiratory pressure
  Interventions: Other: Combined training; Other: Electrical stimulation; Other: Control group
- Control group (No Intervention): No intervention.

INTERVENTIONS:
Other: Combined training — FES will be applied at 15 Hz, 0.4 ms pulse width, 10-s contraction time, 50-s resting time and maximum tolerable intensity, 3 sessions per week, for 12 weeks. The IMT will also be performed for 12 weeks, 5 sessions per week, with an intensity of 30% of maximal inspiratory pressure.
  Other Names: Electric stimulation; Electrical stimulation; Inspiratory muscle training; Breathing exercises
  Arms: Electrical stimulation; Inspiratory muscle training
Other: Electrical stimulation — FES will be applied at 15 Hz, 0.4 ms pulse width, 10-s contraction time, 50-s resting time and maximum tolerable intensity, 3 sessions per week, for 12 weeks
  Other Names: Electric stimulation; Eletric stimulation therapy
  Arms: Combined training; Inspiratory muscle training
Other: Inspiratory muscle training — IMT will be performed for 12 weeks, 5 sessions per week, with an intensity of 30% of maximal inspiratory pressure
  Other Names: Respiratory muscle training; Breathing exercises
  Arms: Combined training; Electrical stimulation
Other: Control group — No intervention
  Arms: Combined training; Electrical stimulation; Inspiratory muscle training

SUMMARY:
The purpose of this study is to assess the effects of functional electrical stimulation associated with inspiratory muscle training on functional capacity and quality of life in heart failure patients.

DETAILED DESCRIPTION:
The aim of this study is to assess the effects of the functional electrical stimulation (FES) associated with inspiratory muscle training (IMT) on functional capacity and quality of life in patients with heart failure (HF). A randomized clinical trial with 60 HF patients (functional class II-IV) will be randomly assigned to the FES, IMT, IMT associated with FES or control group. FES will be applied at 15 Hz, 0.4 ms pulse width, 10-s contraction time, 50-s resting time and maximum tolerable intensity, 3 sessions per week, for 12 weeks. The IMT will also be performed for 12 weeks, 5 sessions per week, with an intensity of 30% of maximal inspiratory pressure. Acute and chronic effects of interventions on functional capacity, quality of life, peripheral muscle strength, pulmonary function, respiratory muscle strength and endurance, endothelial function, autonomic control and oxidative stress will be analyzed in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stable heart failure and New York Heart Association (NYHA) class II-IV
* Aged 30-70 years
* Left ventricular ejection fraction less than 35% determined by echocardiography and optimized pharmacological treatment (unchanged 1 month prior to study)

Exclusion Criteria:

* Patients with unstable heart failure
* NYHA class I
* Unstable angina pectoris and ventricular arrhythmia
* Implanted cardiac pacemaker
* Acute pulmonary diseases
* Chronic renal failure or dialysis
* Acute myocardial infarction 3 months before the inclusion in the study
* Acute inflammatory diseases
* Peripheral vascular disease
* Neurologic disease
* Musculoskeletal pathologies
* Malignancies or being an active smoker

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-03; Primary Completion 2016-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Functional capacity | 12 weeks
  To assess the effects of the functional electrical stimulation (FES) associated with inspiratory muscle training (IMT) on functional capacity.

SECONDARY OUTCOMES:
Quality of life | 12 weeks
  To assess the effects of the functional electrical stimulation (FES) associated with inspiratory muscle training (IMT) on quality of life.
Peripheral muscle strength | 12 weeks
  To assess the effects of the functional electrical stimulation (FES) associated with inspiratory muscle training (IMT) on peripheral muscle strength.
Pulmonary function | 12 weeks
  To assess the effects of the functional electrical stimulation (FES) associated with inspiratory muscle training (IMT) on pulmonary function.
Respiratory muscle strength | 12 weeks
  To assess the effects of the functional electrical stimulation (FES) associated with inspiratory muscle training (IMT) on respiratory muscle strength.
Endothelial function | 12 weeks
  To assess the effects of the functional electrical stimulation (FES) associated with inspiratory muscle training (IMT) on endothelial function.
Autonomic control | 12 weeks
  To assess the effects of the functional electrical stimulation (FES) associated with inspiratory muscle training (IMT) on autonomic control.
Oxidative stress | 12 weeks
  To assess the effects of the functional electrical stimulation (FES) associated with inspiratory muscle training (IMT) on oxidative stress.

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo DM Plentz, PhD, Principal Investigator — Instituto de Cardiologia do Rio Grande do Sul/Fundação Universitária de Cardiologia
Locations (1):
- Instituto de Cardiologia do Rio Grande do Sul/Fundação Universitária de Cardiologia, Porto Alegre, Rio Grande do Sul, Brazil